CLINICAL TRIAL: NCT02115295
Title: Phase II Study of Cladribine Plus Idarubicin Plus Cytarabine (ARAC) in Patients With AML, HR MDS, or Myeloid Blast Phase of CML
Brief Title: Cladribine, Idarubicin, Cytarabine, and Venetoclax in Treating Patients With Acute Myeloid Leukemia, High-Risk Myelodysplastic Syndrome, or Blastic Phase Chronic Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0648; NCI-2014-01103 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0648 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Acute Biphenotypic Leukemia; Acute Myeloid Leukemia; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Blasts 10 Percent or More of Bone Marrow Nucleated Cells; Blasts 10 Percent or More of Peripheral Blood White Cells; de Novo Myelodysplastic Syndrome; Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Acute Myeloid Leukemia; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute; Blast Crisis; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Cladribine; Cytarabine; gilteritinib; Idarubicin; midostaurin; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cladribine, cytarabine, idarubicin) (Experimental): INDUCTION: Patients receive cladribine IV and cytarabine IV over 1-2 hours on days 1-5 and idarubicin IV over 30-60 minutes on days 1-3. Patients with untreated AML and MDS also receive venetoclax PO on days 2-8. AML patients with known FLT3-ITD or FLT3 kinase domain mutations may receive midostaurin PO BID on days 6-19 or gilteritinib PO QD on days 1-14. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive cladribine IV and cytarabine IV over 1-2 hours on days 1-3 and idarubicin IV over 30-60 minutes on days 1-2. Patients with untreated AML and MDS also receive venetoclax PO on days 2-8. AML patients with known FLT3-ITD or FLT3 kinase domain mutations may receive midostaurin PO BID on days 6-19 or gilteritinib PO QD. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Gilteritinib; Drug: Idarubicin; Other: Laboratory Biomarker Analysis; Drug: Midostaurin; Drug: Venetoclax

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Gilteritinib — Given PO
  Other Names: ASP-2215; ASP2215; Xospata
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-demethoxydaunorubicin; 4-DMDR
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Midostaurin — Given PO
  Other Names: CGP 41251; CGP41251; N-Benzoyl-Staurosporine; N-Benzoylstaurosporine; PKC-412; PKC412; Rydapt
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well cladribine, idarubicin, cytarabine, and venetoclax work in patients with acute myeloid leukemia, high-risk myelodysplastic syndrome, or blastic phase chronic myeloid leukemia. Drugs used in chemotherapy, such as cladribine, idarubicin, cytarabine, and venetoclax, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
Primary Objectives:

I. To determine the complete response rate (CR) of cladribine in combination with idarubicin and cytarabine (araC) in patients with acute myeloid leukemia (AML), high risk (HR) myelodysplastic syndrome (MDS), or myeloid blast phase of chronic myeloid leukemia (CML).

Secondary Objectives:

I. To determine the overall response rate (ORR) of cladribine in combination with idarubicin and araC in patients with AML, HR MDS, or myeloid blast phase of CML.

II. To assess overall survival (OS) and event free survival (EFS) of patients treated with cladribine, idarubicin, and araC (cytarabine).

III. To assess the duration of response to the combination in patients with AML, HR MDS, or myeloid blast phase of CML.

IV. To determine the safety and tolerability of the combination in patients with AML, HR MDS, or myeloid blast phase of CML.

Exploratory Objectives:

I. To study and describe the relationship between pretreatment patient/disease characteristics (including AML-associated molecular abnormalities) and outcome.

II. To identify molecular biomarkers predictive of response to therapy.

III. To study and describe the relationship between patient/disease characteristics, use of intrathecal prophylaxis, and incidence of leptomeningeal disease.

IV. To study the trajectories of leukemia mutations and molecular minimal residual disease (MRD) during the therapy.

OUTLINE:

INDUCTION: Patients receive cladribine intravenously (IV) and cytarabine IV over 1-2 hours on days 1-5 and idarubicin IV over 30-60 minutes on days 1-3. Patients with untreated AML and MDS also receive venetoclax orally (PO) on days 2-8. AML patients with known FLT3-ITD or FLT3 kinase domain mutations may receive midostaurin PO twice daily (BID) on days 6-19 or gilteritinib PO once daily (QD) on days 1-14. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive cladribine IV and cytarabine IV over 1-2 hours on days 1-3 and idarubicin IV over 30-60 minutes on days 1-2. Patients with untreated AML and MDS also receive venetoclax PO on days 2-8. AML patients with known FLT3-ITD or FLT3 kinase domain mutations may receive midostaurin PO BID on days 6-19 or gilteritinib PO QD. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of AML, Acute Biphenotypic Leukemia, or high risk MDS (>/= 10% blasts or IPSS >/= intermediate-2) will be eligible. Patients with CML in Myeloid Blast Phase are also eligible.
2. For Frontline cohort (1 or 4): No prior potentially-curative therapy for leukemia. Prior therapy with hydroxyurea, hematopoietic growth factors, azacytidine, decitabine, ATRA, or a total dose of cytarabine up to 2g (for emergency use for stabilization) is allowed. Patients deemed able to receive venetoclax (ie. insurance clearance) will be assigned to Frontline cohort 4. Patients with secondary AMLwho have been treated for their antecedent myeloid neoplasm will be enrolled into the separate Secondary AML cohort.
3. For Salvage cohort: Patients with previously treated, relapsed or refractory AML, Acute Biphenotypic Leukemia, or CML in Myeloid Blast Phase are eligible.
4. Age </= 65 years.
5. Adequate organ function as defined below:

   * liver function (bilirubin < 2mg/dL, AST and/or ALT <3 x ULN - or <5 x ULN if related to leukemic involvement)
   * kidney function (creatinine < 1.5 x ULN ).
   * known cardiac ejection fraction of > or = 45% within the past 6 months
6. ECOG performance status of ≤ 2.
7. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
8. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient is required prior to their enrollment on the protocol.

Exclusion Criteria:

1. Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided.
2. Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patient with documented hypersensitivity to any of the components of the chemotherapy program.
4. Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2014-05-19 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | Up to 12 months
  CR rate will be determined.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 12 months
  ORR will be determined.
Overall survival (OS) | Up to 12 months
  OS will be assessed.
Event-free survival (EFS) | Up to 12 months
  EFS will be assessed.
Duration of response | Up to 12 months
  Duration of response will be assessed.
Incidence of toxicities | Up to 12 months
  Safety and tolerability of cladribine in combination with idarubicin and cytarabine will be determined.

OTHER OUTCOMES:
Use of intrathecal prophylaxis | Up to 12 months
  The relationship between patient/disease characteristics and use of intrathecal prophylaxis will be studied and described.
Incidence of leptomeningeal disease | Up to 12 months
  The relationship between patient/disease characteristics and incidence of leptomeningeal disease will be studied and described.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Goulart H, Jabbour E, Short NJ, Kadia TM, Pemmaraju N, Takahashi K, Ravandi F, Konopleva M, Jain N. A Phase I/II Trial of Ruxolitinib with Chemotherapy for Patients with Relapsed and/or Refractory Philadelphia-like Acute Lymphoblastic Leukemia. Clin Lymphoma Myeloma Leuk. 2025 Nov;25(11):800-807. doi: 10.1016/j.clml.2025.05.013. Epub 2025 May 20. PMID 40500616
- [Derived] Goulart H, Kantarjian H, Borthakur G, Daver N, DiNardo CD, Jabbour E, Pemmaraju N, Alvarado Y, Atluri H, Yilmaz M, Haddad FG, Marx KR, Rausch C, Loghavi S, Jain N, Garcia-Manero G, Ravandi-Kashani F, Kadia TM. Cladribine, idarubicin, and cytarabine (CLIA) for patients with relapsed and/or refractory acute myeloid leukemia: A single-center, single-arm, phase 2 trial. Cancer. 2025 Apr 15;131(8):e35840. doi: 10.1002/cncr.35840. PMID 40193193
- [Derived] Kadia TM, Reville PK, Borthakur G, Yilmaz M, Kornblau S, Alvarado Y, Dinardo CD, Daver N, Jain N, Pemmaraju N, Short N, Wang SA, Tidwell RSS, Islam R, Konopleva M, Garcia-Manero G, Ravandi F, Kantarjian HM. Venetoclax plus intensive chemotherapy with cladribine, idarubicin, and cytarabine in patients with newly diagnosed acute myeloid leukaemia or high-risk myelodysplastic syndrome: a cohort from a single-centre, single-arm, phase 2 trial. Lancet Haematol. 2021 Aug;8(8):e552-e561. doi: 10.1016/S2352-3026(21)00192-7. PMID 34329576
- [Derived] Morita K, Kantarjian HM, Wang F, Yan Y, Bueso-Ramos C, Sasaki K, Issa GC, Wang S, Jorgensen J, Song X, Zhang J, Tippen S, Thornton R, Coyle M, Little L, Gumbs C, Pemmaraju N, Daver N, DiNardo CD, Konopleva M, Andreeff M, Ravandi F, Cortes JE, Kadia T, Jabbour E, Garcia-Manero G, Patel KP, Futreal PA, Takahashi K. Clearance of Somatic Mutations at Remission and the Risk of Relapse in Acute Myeloid Leukemia. J Clin Oncol. 2018 Jun 20;36(18):1788-1797. doi: 10.1200/JCO.2017.77.6757. Epub 2018 Apr 27. PMID 29702001
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org